CLINICAL TRIAL: NCT05033769
Title: AIRE - Assessing ImmunoResponse Post Eribulin: Eribulin and Immunogenicity in Advanced Breast Cancer - a Prospectively Randomized Phase IV Study
Brief Title: Assessing ImmunoResponse Post Eribulin: Eribulin and Immunogenicity in Advanced Breast Cancer
Acronym: AIRE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut fuer Frauengesundheit (Other)
Collaborators: Eisai GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFG-06-2019; 2020-001938-35 (EudraCT Number); AGO-B-049 (Other: AGO-B-ID)
Record Dates: First submitted 2020-06-19; First posted 2021-09-05 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer Female; Neoplasm, Breast; Breast Cancer Metastatic
Keywords: Immunoresponse
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eribulin (Experimental): Arm A. Eribulin 1.23 mg/m^2, administered as an injection on day 1 and 8 q 21d for a maximum of 4 therapy cycles
  Interventions: Drug: Eribulin Injection [Halaven]
- Paclitaxel (Active Comparator): Paclitaxel 80 mg/m^2, administered as an injection on day 1, 8 and 15 q21d for a maximum of 4 therapy cycles
  Interventions: Drug: Paclitaxel injection

INTERVENTIONS:
Drug: Eribulin Injection [Halaven] — on days 1 and 8 q21d
  Other Names: Eribulin
  Arms: Eribulin
Drug: Paclitaxel injection — on days 1, 8, and 15 q21d
  Other Names: Paclitaxel
  Arms: Paclitaxel

SUMMARY:
After progression of disease after one chemotherapy, metastatic breast cancer patients will be randomized 1:1 to one of the following treatment arms:

Arm A. Eribulin Arm B. Paclitaxel

Blood draws for immune analysis will be performed before start of therapy, on day 1 of cycle 2 and on day 21 of cycle 4 (end of therapy) for the primary study aim. Patients will be treated under study conditions for a maximum of 4 therapy cycles.

DETAILED DESCRIPTION:
This is a prospective, randomized Phase IV study. Patients who progressed after one chemotherapy in the metastatic setting will be randomized 1:1 to one of the following treatment arms. Arm A. Eribulin 1.23 mg/m2 on days 1 and 8 q21d Arm B. Paclitaxel 80 mg/m2 on days 1, 8, and 15 q21d Blood draws for immune analysis will be performed before start of therapy on day 1 of cycle 1, on day 1 of cycle 2 (pre dose each) and on day 21 of cycle 4 (end of therapy) and assessed for the primary study aim. Patients will be treated under study conditions for a maximum of 4 therapy cycles.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to beginning of trial specific procedures
* Subject must be female and aged ≥ 18 years on day of signing informed consent
* ECOG 0-1
* Histologically confirmed, HER2 negative breast cancer determined by core biopsy of tumor lesion. Human epidermal growth factor receptor 2 (HER2) negativity is defined as either of the following by local laboratory assessment: In situ hybridization (ISH) non-amplified (ratio ≤ 2.2), or IHC 0 or IHC 1+.
* Indication for chemotherapy
* Previous therapy with one chemotherapy line
* Target lesion (RECIST 1.1)
* Adequate organ function defined as:

Creatinine Clearance > 50 ml/min ANC ≥ 1.5 x 10 3 /μL Thrombocytes > 100 x 10 3 /μL

Exclusion Criteria:

* HER2 positive disease
* Indication for an anti-hormone treatment
* Active infection requiring systemic therapy.
* Active autoimmune disease or other diseases that requires systemic treatment with corticosteroids or immunosuppressive drugs.
* History of primary or acquired immunodeficiency (including allogenic organ transplant).
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
* Severely impaired liver function (Child Pugh C)
* Hypersensitivity to study medication or any of its components
* Neuropathy (PNP) > Grade 2 (CTCAE 5.0)
* Congenital long QT syndrome
* Preexisting concomitant use of strong CYP3A4 and CYP2C8 inhibiting or inducing drugs
* Life expectancy of less than three months
* Pregnancy (contraception is required according tocontraceptive guidance)
* Lactation
* Known history of following infections: Human immunodeficiency virus (HIV), History of acute or chronic Hepatitis B or Hepatitis C
* Has received a live-virus vaccination within 30 days of planned treatment start. Seasonal flu vaccines that do not contain live virus are permitted.
* Does not agree to blood collection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2021-03-11 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
Immune responsivity (IR) | 12 weeks after therapy start
  defined as ≥ 5% of all T cells from peripheral blood are Ki-67 positive after chemotherapy

SECONDARY OUTCOMES:
Overall response after three months | three months after therapy start
  Overall response
Progression free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Progression free survival
Overall survival | From date of randomization until the date of death from any cause, whichever came first, assessed up to 24 months
  Overall survival
Toxicity and safety of eribulin and paclitaxel | Therapy start until 30 days post last dose
  Toxicity and safety of eribulin and paclitaxel
EORTC QLQC30 | Therapy start until therapy end after 4 cycles up to 12 weeks
  Quality of life assessed via EORTC QLQC30

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Fasching, MD, Prof., Study Chair — Department of Gynecology and Obstetrics, Erlangen University Hospital
Locations (2):
- Germany (2):
  - Department of Gynecology, Tübingen University Hospital, Tübingen, Baden-Wurttemberg
  - Department of Gynecology and Obstetrics, Erlangen University Hospital, Erlangen, Bavaria

IPD SHARING:
Plan to Share IPD: No